CLINICAL TRIAL: NCT01170520
Title: The Addition of rTMS to the Therapy of Adolescents That Suffer From Treatment Resistant Depression: An Open Label Study
Brief Title: Repetitive Transcranial Stimulation (rTMS) for Resistant Depression in Adolescents
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HT 4953
Record Dates: First submitted 2010-07-23; First posted 2010-07-27 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Adolescent Depression
Keywords: adolescent resistant depression; repetitive transcranial magnetic stimulation; treatment of resistant adolescent depression

ARMS (1):
- rTMS (Experimental)
  Interventions: Device: repetitive transcranial Stimulation

INTERVENTIONS:
Device: repetitive transcranial Stimulation — rTMS using the figure of 8 magstim for 4 weeks or 20 work days, using 100% threshold to the LDPFC 42 trains per day 4 sec pretrain inter train interval of 30 sec.

SUMMARY:
The investigators hypothesis that repetitive transcranial Stimulation (rTMS) is a safe and effective add-on therapy for resistent depression in adolescent patients.

A group of adolescents suffering from non psychotic major depression that was resistant to at least 2 drug trials and a trail of psychotherapy will be recruited. After an informed consent procedure for both parents and patients, patients will go through a clinical and cognitive evaluation. They will receive a protocol of 4 weeks (20 work days) of rTMS using the figure of 8 magstim coil at 100% threshold, 42 trains of 4 seconds each, intertrain interval of 30 sec to the LDPC, 1680 pulses per day. Then they will be reevaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age 15-18 years old
* Right hand dominant
* Suffering from major depression
* CDRS > 60
* At least 3 months of current depressive episode
* Failed 2 drug trials (or 3 drug trials if trial terminated prematurely due to side effects) and at least 1 course of psychotherapy
* No contraindication for rtms (safety questionnaire)
* No change in pharmacotherapy in the last month

Exclusion Criteria:

* Schizophrenia or psychotic symptoms
* Hypertension
* Epilepsy
* History of major head trauma
* Metal implements in the head
* History of neurosurgery
* History of severe head migraine
* History of hearing loss or sp cochlear transplantation
* Pregnancy
* Current drug abuse
* Unstable medical condition
* History of manic episode
* Current treatment with lithium or tricyclic or tetracyclic antidepressants

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-08; Primary Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Child Depression Rating Scale (CDRS) comparison before after therapy | 4 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Shalvata Mental health Center, Hod HaSharon
  - Shalvata Mental Health Center, Hod HaSharon